CLINICAL TRIAL: NCT00800878
Title: Chronic Kidney Disease in the Pakistani Population
Brief Title: Chronic Kidney Disease in Pakistani Population
Acronym: CKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Tazeen H Jafar, Aga Khan University
Other Study IDs: R03TW007588 (NIH)
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Renal insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
The Indo-Asian developing countries are facing an epidemic of chronic diseases including hypertension, diabetes and chronic kidney disease (CKD). Diagnosis of early CKD is essential for institution of effective and timely prevention of its complications; costly late stage treatment for end stage renal disease is currently an unfeasible option in these populations. GFR estimates of kidney function provide a common reference standard for all people and are therefore readily applicable by physicians and understood by patients. However, the existing GFR equations yield widely discrepant results in the Indo Asian population, and none of the currently available estimating equations have been validated in this population.

The main objective is to develop a tool which can be used for screening subjects at high risk for developing CKD (with hypertension and diabetes) as well as the general population.

DETAILED DESCRIPTION:
The proposed study is being conducted at the Aga Khan University in collaboration with Tufts-New England Medical Center and Imperial College, UK. It is a population based cross-sectional study using a 2-stage cluster design. The study would be performed on 650 adult subjects from the general population in Karachi.

A new GFR equation specific to a Pakistani population would be developed and validated using the gold standard of measured Insulin GFR. The performance of the new equation will be compared to the existing ones developed in other populations with respect to bias, precision, and accuracy.

The project is likely to contribute significantly to moving the field to kidney disease forward, and its results are likely to have far reaching implications for understanding of CKD and, ultimately, its prevention in Indo-Pakistani populations worldwide.

ELIGIBILITY:
Inclusion Criteria:

* All individuals aged 40 years and above

Exclusion Criteria:

* Shortness of breath on minimal to moderate exertion
* Acute fibril illness
* Doctor diagnosed liver disease
* Doctor diagnosed rheumatological disease
* Heart attack within past three months
* Pregnancy
* Mentally incompetent to give informed consent
* Too frail to travel to clinic
* Bed ridden subjects

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals aged aged 40 years and above in a representative sample of Karachi Demographic Survey constituted the sampling frame. Individuals were screened for hypertension and diabetes and the final sample of about 650 subjects will be randomly selected
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
GFR will be measured as the mean of at least two urinary clearance periods of Inulin

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan